CLINICAL TRIAL: NCT04972344
Title: Preoperative Ionized Magnesium Assessment in Adults: an Observational Study on the Prevalence of Hypomagnesemia
Brief Title: Preoperative Ionized Magnesium Assessment
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, HJ Shin, Associate Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2106-688-304
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Magnesium Deficiency
MeSH Terms: conditions — Magnesium Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ionized magnesium — Assessment of ionized magnesium level

SUMMARY:
The reported incidence of hypomagnesemia is approximately 2% in the general population. Hypomagnesemia is a common problem, occurring in nearly 10%of general hospitalized patients and 17% of hospitalized cancer patients. A higher incidence, up to 60% to 65%, has been found among intensive care unit patients. Hypomagnesemia can potentially cause fatal complications including ventricular arrhythmia, coronary artery spasm, and sudden death. It also associates with increased mortality and prolonged hospitalization.

Magnesium exists in three different forms in the body. In serum, 5-14% of the magnesium is reported to be complexed with anions such as phosphate, bicarbonate, and citrate, 19-33% is reported to be protein-bound (mainly to albumin), and 55-67% is found in the free ionized fraction. Because the amount of bound or complexed Mg can vary significantly, especially in illness, the ionized magnesium can vary in an unpredictable way. Conventional laboratory testing typically only measures total serum magnesium, which is often not reflective of ionized magnesium. Unlike ionized calcium, which is commonly measured and is also readily calculated from the total calcium and albumin levels, ionized magnesium is neither commonly measured nor easily calculated. One study reported that the level of ionized magnesium cannot be predicted by analysis of total magnesium and that the levels of ionized magnesium vary upon different pathophysiological conditions and between individuals. Furthermore, measurement of ionized magnesium in serum might be of great impact in patients for whom magnesium status is required, and the correlation of ionized magnesium and total magnesium is weak in patients for whom magnesium status is required as a whole, and this is the reason why the ionized magnesium should be measured directly.

To date, most of the clinical studies were evaluate the effect of hypomagnesemia on the outcome after surgery using the levels of total serum magnesium. However, the portion of extracellular magnesium that is physiologically active is in the various process is ionized magnesium. So, it is important to evaluate the level of ionized magnesium in surgical patients to predict the outcomes after surgery. Unfortunately, clinical trial regarding the effect of the concentrations of ionized magnesium on the surgical patients is limited.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery
* Aged ≥ 19
* Fasted ≥ 8 hours

Exclusion Criteria:

* Chronic kidney disease
* Aged < 19
* Fasted < 8 hours
* Patients who were taking magnesium

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 536 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Ionized magnesium | within 10 minutes after induction of anesthesia; 10 minutes before the end of surgery
  Assess the ionized magnesium level

SECONDARY OUTCOMES:
total magnesium | within 10 minutes after induction of anesthesia
  Assess the total magnesium level

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Jung Shin, MD., PhD., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No